CLINICAL TRIAL: NCT00763555
Title: A Multicenter, Randomized, Vehicle-controlled, Efficacy and Safety Study of CD2027 3µg/g Oily Spray Applied Twice Daily for 8 Weeks in Subjects With Plaque-type Psoriasis
Brief Title: Efficacy and Safety Study of CD 2027 Spray in Subjects With Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18119
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Results first posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-04

CONDITIONS: Psoriasis
Keywords: psoriasis; spray; calcitriol
MeSH Terms: conditions — Psoriasis | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Calcitriol 3 mcg/g Spray (Experimental)
  Interventions: Drug: CD 2027
- Calcitriol Vehicle (Placebo Comparator)
  Interventions: Drug: Calcitriol Vehicle

INTERVENTIONS:
Drug: CD 2027 — Participants applied Calcitriol 3 mcg/g spray topically to the affected areas twice daily for 8 weeks.
  Other Names: Calcitriol
  Arms: Calcitriol 3 mcg/g Spray
Drug: Calcitriol Vehicle — Participants applied placebo matched to Calcitriol 3 mcg/g spray topically to the affected areas twice daily for 8 weeks.
  Arms: Calcitriol Vehicle

SUMMARY:
This was a multicenter, randomized, vehicle-controlled, double-blind parallel group study to evaluate the efficacy and safety of CD 2027 Oily Spray applied twice daily for 8 weeks in participants with plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of plaque-type psoriasis up to 20% of body surface area (BSA) involved excluding the scalp, with a Global Severity Score of at least 3 (moderate) at Screening
* Participant presents with a representative target lesion that is at least 16 cm² in area, is located on the non-bony areas of the skin, has a Scaling Score up to 2 (moderate), has a DSS of at least 4

Exclusion Criteria:

* Other type of psoriasis (other than plaque)
* Significant abnormal lab findings
* Hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Tennessee Clinical Research Center, Nashville, Tennessee
- Canada (4):
  - Stratica Medical, Edmonton, Alberta
  - Ultranova Skincare, Barrie, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - K. Papp Clinical Research, Inc., Waterloo, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in United States and Canada between 22 September 2008 and 23 January 2009.
Pre-assignment Details: A total of 111 participants were screened in the study. Out of which, 88 participants were randomized to receive Calcitriol 3 micrograms per gram (mcg/g) spray or its vehicle.
Groups:
- Calcitriol 3 mcg/g Spray: Participants applied Calcitriol 3 mcg/g spray topically to the affected areas twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Started | 44 | 44
Completed | 40 | 34
Not Completed | 4 | 10
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population is defined as all participants who were randomized and to whom medication is dispensed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 36 | 77
  >=65 years | 3 | 8 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 24 | 32 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 42 | 40 | 82
  Black | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success Rate 1 (SR1) at Week 8
Description: Success Rate 1 was defined as percentage of participants who achieved at least 2-grade improvement from Baseline on Global Severity Score (GSS) at Week 8. GSS is a 5-point scale which ranges from 0-4, where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe, higher score indicated higher severity. All missing values were imputed by last observation carried forward (LOCF).
Time Frame: Week 8
Population: ITT population is defined as all participants who were randomized and to whom medication is dispensed.
Measure: Number; unit: percentage of participants
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 44 | 44
percentage of participants | 4.5 | 0.0

2. Primary Outcome: Percentage of Participants With Success Rate 2 (SR2) at Week 8
Description: Success Rate 2 was defined as percentage of participants who achieved "clear" or "almost clear" on GSS at Week 8. GSS is a 5-point scale which ranges from 0-4, where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe, higher score indicated higher severity. All missing values were imputed by last observation carried forward (LOCF).
Time Frame: Week 8
Population: ITT population is defined as all participants who were randomized and to whom medication is dispensed.
Measure: Number; unit: percentage of participants
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 44 | 44
percentage of participants | 4.5 | 0.0

3. Primary Outcome: Change From Baseline in Dermatologic Sum Score (DSS) at Week 8
Description: DSS is the sum of all the individual score of evaluated target lesion that includes plaque elevation (abnormal thickness of the psoriasis lesion), erythema (abnormal redness of the skin), and scaling (shedding of the stratum corneum). Each individual parameters evaluated the affected area by using a 5-point scale ranging from 0 to 4, that is, 0 = None; 1 = Mild; 2 = Moderate; 3 = Severe and 4 =Very severe, where higher score indicated worst condition. All missing values were imputed by last observation carried forward (LOCF). The total score of each parameter ranges from 0-12, where higher score indicated worst condition.
Time Frame: Baseline, Week 8
Population: ITT population is defined as all participants who were randomized and to whom medication is dispensed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 44 | 44
score on a scale | -1.2 (1.66) | -1.0 (1.55)

4. Primary Outcome: Percentage of Participants With at Least 1-Grade Improvement From Baseline in Erythema, Scaling and Plaque Elevation
Description: Erythema (abnormal redness of skin) score is a 5-point scale: 0=None (No detectable erythema. Skin of normal color); 1=Mild (Slight pinkness present); 2=Moderate (Definite redness, easily recognized); 3=Severe (Intense redness) and 4=Severe (Very Intense redness). Scaling (shedding of stratum corneum) score is a 5- point scale: 0=None (No shedding); 1=Mild (Barely perceptible shedding, noticeable only on light scratching or rubbing); 2=Moderate (Obvious but not profuse shedding); 3=Severe (heavy scale production) and 4=Very severe (very thick scales). Plaque elevation (abnormal thickness of psoriasis lesion) score was a 5- point scale: 0=None (Normal skin thickness. No elevation of skin); 1=Mild (Barely perceptible elevation (by touching) of psoriasis plaques); 2=Moderate (Obvious elevation above normal skin level; moderate thickening); 3=Severe (definite thick elevation above normal skin level) and 4=Severe (Very thick elevation).
Time Frame: Baseline, Week 8
Population: ITT population is defined as all participants who were randomized and to whom medication is dispensed.
Measure: Number; unit: percentage of participants
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 44 | 44
percentage of participants
  Erythema | 38.6 | 25.0
  Scaling | 40.9 | 36.4
  Plaque elevation | 34.1 | 36.4

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily had a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: up to Week 8
Population: The Safety population is defined as all participants in the ITT population who have applied the study medication at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 44 | 44
Participants | 11 | 9

6. Secondary Outcome: Percentage of Participants With a Local Tolerability Score Worse Than Baseline Score
Description: Local tolerability skin assessments were performed by the investigator and based on 5-point scale which ranges from 0 to 4. 0 = none (no evidence of local intolerance); 1=mild (minimal erythema and/or edema, slight glazed appearance); 2 = moderate (definite erythema and/or edema with peeling and/or cracking but needs no adaptation of posology); 3 = severe (erythema, edema glazing with fissures, few vesicles or papules) and 4 = very severe (strong reaction spreading beyond the treated area, bullous reaction, erosions). Higher grades indicated worsening of condition. Percentage of participants with increase in score by Week 8 from baseline has been presented here, where the row titles indicate participant's new scores by Week 8.
Time Frame: up to Week 8
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 44 | 44
percentage of participants
  1 = mild | 4.5 | 7.0
  2 = moderate | 2.3 | 0.0
  3 = severe | 2.3 | 4.7
  4 = very severe | 2.3 | 2.3

7. Secondary Outcome: Change From Baseline in Calcitriol Plasma Levels
Description: Change from baseline in calcitriol plasma levels were reported.
Time Frame: Baseline, Week 8
Population: The Safety population is defined as all participants in the ITT population who have applied the study medication at least once. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
picograms per milliliter (pg/mL) | -2.89 (23.971) | -8.82 (22.873)

8. Secondary Outcome: Change From Baseline in Serum Calcium Homeostasis Parameter: Albumin
Description: Change from baseline in serum calcium homeostasis parameter (Albumin) were reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
grams per deciliter (g/dL) | -0.16 (0.253) | -0.08 (0.230)

9. Secondary Outcome: Change From Baseline in Serum Calcium Homeostasis Parameter: Albumin-adjusted Calcium
Description: Change from baseline in serum calcium homeostasis parameter (Albumin-adjusted calcium) were reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
milligrams per deciliter (mg/dL) | 0.07 (0.310) | 0.03 (0.262)

10. Secondary Outcome: Change From Baseline in Serum Calcium Homeostasis Parameter: Calcium
Description: Change from baseline in serum calcium homeostasis parameter (Calcium) were reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
mg/dL | -0.09 (0.283) | -0.05 (0.328)

11. Secondary Outcome: Change From Baseline in Serum Calcium Homeostasis Parameter: Phosphorus
Description: Change from baseline in serum calcium homeostasis parameter (Phosphorus) were reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
mg/dL | -0.07 (0.437) | 0.02 (0.535)

12. Secondary Outcome: Change From Baseline in Serum Calcium Homeostasis Parameter: Parathyroid Hormone (PTH) Intact
Description: Change from baseline in serum calcium homeostasis parameter (PTH intact) were reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
pg/mL | 7.16 (25.215) | 5.15 (18.480)

13. Secondary Outcome: Change From Baseline in Blood Chemistry: Alkaline Phosphatase, Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT)
Description: Change from baseline in Blood Chemistry: Alkaline Phosphatase, AST and ALT were reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
international units per liter (IU/L)
  Alkaline Phosphatase | 0.58 (8.362) | -1.03 (17.150)
  AST | 1.42 (9.014) | -0.35 (8.110)
  ALT | 0.72 (8.564) | -1.75 (11.151)

14. Secondary Outcome: Change From Baseline in Blood Chemistry: Bilirubin Direct, Bilirubin Total, Blood Urea Nitrogen (BUN) and Creatinine
Description: Change from baseline in Blood Chemistry: Bilirubin Direct, Bilirubin Total, BUN and Creatinine were reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 43 | 40
mg/dL
  Bilirubin Direct | -0.02 (0.048) | -0.03 (0.054)
  Bilirubin Total | 0.01 (0.208) | 0.03 (0.200)
  BUN | 0.65 (3.592) | 0.55 (3.250)
  Creatinine | -0.01 (0.130) | 0.03 (0.103)

15. Secondary Outcome: Change From Baseline in Vital Sign Parameter: Heart Rate
Description: Change from baseline in vital sign parameter: heart rate was reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 40 | 34
beats per minute | 3.1 (7.63) | 1.4 (8.53)

16. Secondary Outcome: Change From Baseline in Vital Sign Parameter: Systolic Blood Pressure and Diastolic Blood Pressure
Description: Change from baseline in vital sign parameter: Systolic Blood Pressure and Diastolic Blood Pressure was reported.
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
Number analyzed (Participants) | 40 | 34
millimeter of mercury (mmHg)
  Systolic Blood Pressure | 0.7 (14.03) | -1.4 (11.01)
  Diastolic Blood Pressure | 0.2 (7.43) | -1.0 (8.54)

ADVERSE EVENTS:
Time Frame: up to Week 8
Description: The Safety population is defined as all participants in the ITT population who have applied the study medication at least once.
Arm/Group | Calcitriol 3 mcg/g Spray | Calcitriol Vehicle
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/44
Other Adverse Events (participants affected / at risk) | 10/44 | 8/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcitriol 3 mcg/g Spray (N=44) | Calcitriol Vehicle (N=44)
Coronary artery disease (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcitriol 3 mcg/g Spray (N=44) | Calcitriol Vehicle (N=44)
Nasopharyngitis (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Blood calcium increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other